CLINICAL TRIAL: NCT00145483
Title: A Multicentre, Double-Blind, Randomized, Placebo-Controlled, Parallel Group Study Of The Efficacy and Safety Of Sildenafil Given For The Acute Treatment Of Meniere's Disease
Brief Title: Sildenafil For Meniere's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1481107
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Meniere's Disease
MeSH Terms: conditions — Meniere Disease | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: Sildenafil

SUMMARY:
Meniere's disease affects a person's sense of balance. An attack can last 20 minutes to 2 hours or longer. Symptoms include rotational vertigo, hearing loss, tinnitus and a sensation of fullness in the affected ear and may be associated with nausea and vomiting. One hypothesis is that Meniere's disease is caused by the excessive accumulation of fluid in the balance tubes within the inner ear. Sildenafil may alleviate the symptoms due to its vasodilatory activity. The purpose of this study is to assess the safety and efficacy of sildenafil (Viagra) compared with placebo on symptoms during one acute attack.

ELIGIBILITY:
Inclusion Criteria:

* Active Meniere's disease (2 or more definitive spontaneous episodes of vertigo 20 minutes or longer, plus hearing loss on at least 1 occasion, tinnitus or aural fullness) with confirmed diagnosis

Exclusion Criteria:

* Pregnant or breast feeding females or fertile females unwilling to use agreed contraceptive methods
* severe Meniere's diseased (more than 8 attacks per month)
* previous ear surgery
* intratympanic perfusions of steroids or gentamicin; requiring other medications contraindicated for Viagra (eg. nitrates)
* with medical conditions that make Viagra contraindicated

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2002-06-18 (Actual); Primary Completion 2006-11-08 (Actual); Study Completion 2006-11-08 (Actual)

PRIMARY OUTCOMES:
Vertigo Response (4 x 6 point scale); Balance (6 point scale)

SECONDARY OUTCOMES:
Hearing/Tinnitus; Ear, Nose & Pressure/Fullness; Perf. daily activities; Nausea; Vomiting; Func. Response; Duration of the Attack and Vertigo; Rescue Medications Use; Acceptability to subject; Composite Assessment Score; Comparison to Previous Attack

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Australia (4):
  - Pfizer Investigational Site, Bondi Junction, New South Wales
  - Pfizer Investigational Site, Brisbane, Queensland
  - Pfizer Investigational Site, East Melbourne, Victoria
  - Pfizer Investigational Site, Melbourne, Victoria

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481107&StudyName=Sildenafil+For+Meniere%27s+Disease+